CLINICAL TRIAL: NCT05322096
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center, Phase 2 Study to Evaluate Efficacy, Safety, and Tolerability of RGH-706 in Prader-Willi Syndrome
Brief Title: Study to Evaluate Efficacy, Safety, and Tolerability of RGH-706 in Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-706-003; 2021-004262-35 (EudraCT Number)
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi Syndrome; Obesity; Hyperphagia control
MeSH Terms: conditions — Prader-Willi Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RGH-706 (Experimental): Dose A once daily for 6 weeks
  Interventions: Drug: RGH-706
- Placebo (Placebo Comparator): Placebo once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGH-706 — Capsules
  Oral administration
  Arms: RGH-706
Drug: Placebo — Capsules
  Oral administration
  Arms: Placebo

SUMMARY:
RGH-706 is a novel, potent, and orally active MCHR1 antagonist drug candidate discovered and being developed by Gedeon Richter Plc. for weight management.

This will be the first Phase 2, proof-of-concept study using RGH-706 and is the third study in the clinical development program for RGH-706. The aim of this study is to evaluate the efficacy, safety, and tolerability of RGH-706 in patients with Prader-Willi Syndrome (PWS).

ELIGIBILITY:
Age Limits:

* In United States (USA), minimum age will be 17 years old.
* In European Union (EU) countries, minimum age will be 18 years old.

Inclusion Criteria:

* Male or female patients aged ≥17 years in USA at screening or aged ≥18 years in EU at screening
* Genetically confirmed diagnosis of PWS
* HQ-CT total score ≥14 at screening
* Body weight ≥40 kg/88 lbs and ≤200 kg/450 lbs
* Stable body weight
* Negative pregnancy test for females of childbearing potential and nonlactating at screening.
* Patients must be able to provide or have a parent or guardian who is able to provide written informed consent and/or assent (as applicable)
* Patients must have at least 1 consistent and reliable primary caregiver

Exclusion Criteria:

* Severe psychiatric disorders (eg, schizophrenia, bipolar disorder, or major depressive disorder), recent (within 6 months)
* Risk of suicide according to the investigator's judgment
* Uncontrollable diabetes mellitus or diabetes mellitus requiring insulin administration
* Poorly controlled hypothyroidism or hyperthyroidism
* Chronic or acute liver disease
* History of bariatric surgery procedure
* Uncontrolled obstructive sleep apnea.
* History of malignancy within 5 years of screening
* Systolic blood pressure (BP) ≥160 mmHg and/or diastolic BP ≥100 mmHg, pulse rate ≥100/min at screening.
* Use of weight-lowering pharmacotherapy within 6 months prior to screening.
* Known QT prolongation
* Clinically relevant laboratory abnormalities
* Any other condition that, in the investigator's opinion, might indicate that the patient is unsuitable for the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
There are no Primary Outcome Measures | There are no Primary Outcome Measures

OTHER OUTCOMES:
Change from baseline in the 9-item Hyperphagia Questionnaire for Clinical Trials (HQ-CT) | Baseline to Day 42
  The HQ-CT is a questionnaire designed to measure symptoms of food-related preoccupations, problems, and behaviors completed by the caregiver. The scale provides a composite value from 9 questions, each rated on a scale of 0 to 4 units (possible total score range: 0 to 36).
  Higher scores represent increased hyperphagia.
Change from baseline in the 9-item Hyperphagia Questionnaire for Clinical Trials (HQ-CT) | Baseline to Days 28, 56, 98 and 133
  The HQ-CT is a questionnaire designed to measure symptoms of food-related preoccupations, problems, and behaviors completed by the caregiver. It consists of 9 items, with a 2-week recall period. The scale provides a composite value from 9 questions, each rated on a scale of 0 to 4 units (possible total score range: 0 to 36). Higher scores represent increased hyperphagia.
Change from baseline in Hyperphagia Questionnaire for Clinical Trials (HQ-CT) domain scores (drive and severity, self-directed behavior) | Baseline to Days 28, 42, 56, 98 and 133
  The HQ-CT is a questionnaire designed to measure symptoms of food-related preoccupations, problems, and behaviors completed by the caregiver. The scale provides a composite value from 9 questions, each rated on a scale of 0 to 4 units (possible total score range: 0 to 36). Higher scores represent increased hyperphagia.
Absolute change from baseline in body weight | Screening, Days 1, 14, 28, 42, 56, 98 and 133
Percentage change from baseline in body weight | Screening, Days 1, 14, 28, 42, 56, 98 and 133
Change from baseline in waist circumference | Screening, Days 1, 14, 28, 42, 56, 98 and 133
Change from baseline in body mass index (BMI) | Screening, Days 1, 14, 28, 42, 56, 98 and 133
Change from baseline in metabolic biomarkers measured from serum | Baseline to Day 42
Change from baseline in Clinical Global Impression-Severity (CGI-S) | Baseline to Days 28, 42 and 56
  The CGI-S rates overall symptom severity on a 4-point scale ranging from 1 (normal) to 7 (severely symptomatic), as assessed by the investigator.
Clinical Global Impression-Improvement (CGI-I) | Days 28 and 42
  The CGI-I is a single statement designed to assess the investigator's overall perception of change in the patient's condition across the course of the clinical trial. The CGI-I uses a 7-point response scale ranging from 1 (very much improved) to 7 (very much worse).
Change from baseline in Caregiver Global Impression-Severity (CaGI-S) | Baseline to Days 2 and 42
  The CaGI-S rates severity of the patient's food-related behavior assessed by the caregiver following a 4-point scale ranging from 0 (none) to 3 (severe).
Caregiver Global Impression-Change (CaGI-C) | Days 28, 42, 56, 98 and 133
  The CaGI-C is a single item designed to assess the primary caregiver's overall perception of change in the patient's hyperphagia symptoms. Responses are rated using a 7-point scale ranging from 1 (much better) to 7 (much worse).
Change from baseline in Zarit Burden Interview-22 (ZBI-22) | Baseline to Day 42
  The ZBI-22 is a self-reported questionnaire in which primary caregivers rate the level of burden currently experienced while taking care of the patient rated on a 5-point scale ranging from 0 (never) to 4 (nearly always).
Safety - Incidence of treatment-emergent adverse events (TEAEs) | Screening thru study end; Up to 24 weeks
Safety - Incidence of clinically significant findings in laboratory values | Screening thru study end; Up to 24 weeks
  Clinical laboratory evaluations (hematology, clinical chemistry, coagulation and lipids, thyroid function test, and urinalysis)
Safety - Incidence of clinically significant findings in vital signs | Screening thru study end; Up to 24 weeks
  Vital signs measurements (body temperature, pulse rate, respiration rate, blood pressure [BP])
Safety - Incidence of clinically significant findings in 12-lead electrocardiograms (ECGs) | Screening thru study end; Up to 24 weeks
Safety - Incidence of clinically significant findings in Columbia-Suicide Severity Rating Scale (C-SSRS) | Screening thru study end; Up to 24 weeks
  The C-SSRS is a clinician-rated instrument that captures the occurrence, severity, and frequency of suicidal ideation and/or behavior during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if suicidal ideation and/or behavior occurred.
Safety - Incidence of clinically significant findings in laboratory values physical examinations | Screening thru study end; Up to 24 weeks
PK Cohort - Individual plasma concentrations of RGH-706 and its metabolite desisopropyl RGH-706 maximum observed plasma concentration (Cmax) | Days 14, 42, 43, 44 and 46
PK Cohort - Individual plasma concentrations of RGH-706 and its metabolite desisopropyl RGH-706 time of the maximum observed plasma concentration (Tmax) | Days 14, 42, 43, 44 and 46
PK Cohort - Individual plasma concentrations of RGH-706 and its metabolite desisopropyl RGH-706 area under the plasma concentration-time curve to the end of the dosing period (AUC0-24) | Days 14, 42, 43, 44 and 46
PK Cohort - Individual plasma concentrations of RGH-706 and its metabolite desisopropyl RGH-706 minimum observed plasma concentration (Cmin) | Days 14, 42, 43, 44 and 46
PK Cohort - Individual plasma concentrations of RGH-706 and its metabolite desisopropyl RGH-706 accumulation ratio (Rac) | Days 14, 42, 43, 44 and 46

CONTACTS AND LOCATIONS:
Locations (23):
- United States (6):
  - Rady Children's Hospital-San Diego, San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Langone Hospital-Long Island, Mineola, New York
  - Morgan Stanley Children's Hospital of NewYork-Presbyterian, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
- General University Hospital, Prague, Czechia
- France (3):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hôpital Larrey, Toulouse
- Italy (6):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Giannina Gaslini, Genova
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù, Roma
  - Oasi Maria SS, Troina
- Spain (7):
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital General Universitario Gregorio Maranon-Instituto Provincial de Psiquiatria y Salud Mental, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Parc Taulí Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No